## Impact of Beef on Metabolites and Inflammation

Dr. Mary Miles

NCT #: 05460754

July 13, 2022

## Statistical Analysis:

Analysis of blood markers and amino acids will be done in the latest version of R available at the time. Paired t-tests will be used to assess baseline anthropometrics between groups to identify any possible covariates to account for. Fasting blood markers and amino acids will also be assessed with paired t-tests to determine any baseline differences in participants that may impact the postprandial results. Net area under the curve (AUC) will be calculated in R for all postprandial markers. The AUC values form each condition will be compared via paired t-tests. Repeated measures ANOVA will be used to assess differences throughout the 4-hour time course for all postprandial markers.